CLINICAL TRIAL: NCT06718907
Title: Mitigating Response to Stressors in the Pregnant Woman
Brief Title: Mitigating Response to Stressors in Pregnant Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NSU 2023-231
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Pregnancy
Keywords: stressors, chronic stress, pregnancy, stress regulation, stress management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stress Exposure and Management (Experimental): All pregnant participants will be exposed to a 50 second-mild stressful stimulus and a 50 second- relaxant to record physiological responses. The participants will then independently practice easy stress management techniques at home, such as breathing and listening to music. They will do so for one week after the initial data collection.
  Interventions: Behavioral: Simulated stimuli; Behavioral: Stress Management

INTERVENTIONS:
Behavioral: Simulated stimuli — Participants will be exposed to a video stimuli in order to assess biophysiological and physiological responses to the stressor and relaxant.
Behavioral: Stress Management — Participants will practice stress management and stress reduction at home, independently.

SUMMARY:
Stress-induced pregnancy complications are significant contributors to preterm labor as well as maternal and perinatal morbidity and mortality. The goals of this study are two folds: first it aims to capture the pregnant woman's journey to seek and receive prenatal care. Second, this study aims to develop models that 1) assess the adverse health and biological effects of social factors on pregnant women who experience repeated or chronic stress, 2) address how stress can be mitigated in pregnant women from different backgrounds who experience high stress.

DETAILED DESCRIPTION:
Maternal stress-induced complications are correlated with gestational hypertension, infant low birth weight, and developmental disruption. Various social determinants of health are contributors to stress in pregnant women; factors such as socioeconomic status, education, access to prenatal care, and neighborhood conditions are some of the most identified psychosocial causes of prenatal stress. Further, chronic psychosocial stress is identified as a significant contributor to biophysiological damages such as accelerated telomere shortening in the mother as well as the offspring. Using a public health approach, this research study proposes to gather evidence to assess how response to stress is modulated and how it is captured in and affects pregnant women, with history of prolonged exposure to harmful stressors. More relevant to this study, individuals who have repeated exposure to stressors have poorly managed response to stress and display frequent elevated heart rates due to biological and physiological disruptions. Evidence from the literature suggests that having a support system and utilizing stress management techniques moderate and buffer the effects of stress on physiological measures while facilitating emotional recovery.

ELIGIBILITY:
Inclusion Criteria: in 24 weeks gestation or more

* between 21 and 37 years of age

Exclusion Criteria:

* in less than 24 weeks gestation
* high risk pregnancies

Ages: 21 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 50 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Stress level change | 4-8 weeks
  change in stress measures as assessed by salivary cortisol levels from collected saliva before and after practicing stress management techniques. Cortisol levels are measured in ug/dL.

CONTACTS AND LOCATIONS:
Overall Officials: Gesulla Cavanaugh, PhD, MPH, MS, Principal Investigator — Nova Southeastern University
Locations (1):
- Nova Southeastern University, Davie, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Working with vulnerable populations and possible individuals from clinics located in underserved communities.